CLINICAL TRIAL: NCT04120545
Title: Effectiveness of Microcurrents Therapy in Overactive Bladder : Controlled and Randomized Triple Blind Clinical Trial
Brief Title: Effectiveness of Microcurrents Therapy in Overactive Bladder.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Las Palmas de Gran Canaria (Other)
Responsible Party: Principal Investigator, Aníbal Báez Suárez, Clinical Professor, University of Las Palmas de Gran Canaria
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NESAob
Record Dates: First submitted 2019-10-06; First posted 2019-10-09 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Overactive Bladder; Urinary Incontinence
Keywords: physical therapy modality; Electric Stimulation Therapy; Urologic Diseases; Pelvic Floor Disorders
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence; Urologic Diseases; Pelvic Floor Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microcurrents (Experimental): Intervention with microcurrents: application of 6 electrodes per extremity and an adhesive electrode at C7, L3 or S1 level depending on the session number.
  Interventions: Device: Microcurrents
- Placebo microcurrents (Placebo Comparator): Intervention with microcurrents: application of 6 electrodes per extremity and an adhesive electrode at C7, L3 or S1 level depending on the session number.
  Interventions: Device: Placebo Microcurrents

INTERVENTIONS:
Device: Microcurrents — The electrodes will be placed with the help of gloves and adapted socks for 1 hour, twice a week, until 10 intervention sessions are completed. In addition, depending on the session, an adhesive electrode will be placed at the level of C7, L3 or S1.
  Characteristics of microcurrents: pulsed monophasic rectangular wave with a pulse of 1.3 s and pause of 300 ms, voltage 3 mV and intensity 0.5 μA.
  Arms: Microcurrents
Device: Placebo Microcurrents — The same protocol described for the experimental group will be applied, but microcurrents device which will be previously manipulated and tested with an oscilloscope so that they do not emit electrical currents
  Arms: Placebo microcurrents

SUMMARY:
The purpose of this study is to investigate the effect on the overactive bladder in women using a care protocol plus the application of microcurrent patches during 1 hours per session compared to the effect of the same protocol plus placebo electric stimulation.

DETAILED DESCRIPTION:
The design of this study is a multicentric, parallel, randomised, triple blind clinical trial with placebo control.

The size of the sample will be 56 participants who come to referral hospitals. They will be randomized in two groups: control or experimental.

The variables of the study will be collected at three time points: before the intervention, during the intervention and at the end of the intervention.

The statistical analysis will be an intention-to-treat analysis. For the main outcomes variables a two factor ANOVA will-be performed (intervention-time) with a post-hoc analysis with kruskal wallis correction correction. Statistical significance will be defined as p <0.05

ELIGIBILITY:
Inclusion Criteria:

* Women, over 18 years of age and with urinary incontinence (3 or more times per week) or overactive bladder (8 or more emptied per day, and / or 2 or more at night) who have received, or not, active / alternative treatment for this pathology.
* Under competent cognitive conditions to participate in the study and trained to complete the study questionnaires.
* Without contraindications for a treatment with microcurrents: Pacemakers, pregnant women, internal bleeding, do not apply electrodes on skin in poor condition, with ulcerations or wounds, acute febrile processes, acute thrombophlebitis and / or electricity phobia.

Exclusion Criteria:

* People with lifestyle habits (diet, amount of fluid ingested) extreme or singular (eg person who consumes 5 liters of water a day).
* Presence of urinary fistula.
* Men. Men will be excluded to avoid the potential influence of prostate problems, the main causes of the symptoms described.
* Urinary tract infection, or relapses: 5 or more infections in the last 12 months.
* Participants with bladder stones.
* Hematuria during the trial period.
* Pregnancy or plans for it during the study.
* The patient has had a hysterectomy.
* Pathology of the central or peripheral nervous system.
* Diabetes without controlled and guaranteed medical treatment its stabilization.
* Diabetes that affects the peripheral nerves.
* Treated with anticoagulant.
* Current use of anticholinergics and beta adrenergic use in the last 4 weeks.
* Currently treated with botox injections for the bladder or in the last year.
* Current treatment with interstim or interstim device currently implanted.
* Obstruction of the bladder outlet.
* Urinary retention.
* Painful bladder syndrome / interstitial cystitis.
* Treatment with more than two antidepressants and / or multiple benzodiazepines, as well as anti-epileptics.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men will be excluded to avoid the potential influence of prostate problems, the main causes of the symptoms described.
Enrollment: 56 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-12-04 (Actual)

PRIMARY OUTCOMES:
Urinary Incontinence | Through study completion, an average of 1 year
  The reduction of at least 25% urination will be considered successful. This result is measured objectively from the voiding diary.

SECONDARY OUTCOMES:
Urinary Incontinence II | Between the first and the fourth week of intervention.
  Change in the number of urination / day compared to baseline, at the fourth week.
Urinary Incontinence III | Between the fourth and the eighth week of intervention.
  Change in the number of urinary incontinence episodes / day at 4 weeks and 8.
Nocturia | Average number of nocturia episodes measured in a diary of 3 days before each visit.
  Change in the number of nocturia episodes every 24 hours
Bladder Control Self-Assessment Hyperactive | After 5 weeks of intervention.
  Changes in the value of the Hyperactive Bladder Control Self-Assessment Questionnaire
International Consultation on Incontinence questionnaire | It will be completed at the beginning of the study, at week 4 and at 8 of the treatment
  It is a questionnaire in which the experience is answered daily individual urination and incontinence
Spanish Short Version of the Functional Outcomes of Sleep Questionnaire (FOSQ-10SV). | Through study completion, an average of 1 year
  This questionnaire measures the impact of daily sleep in daily activity
Quality of life II ( EuroQol-5D) | Through study completion, an average of 1 year
  The main problems or difficulties are collected by patients in 5 dimensions (mobility, self-care, daily activities, pain / discomfort level and anxiety / depression level).

OTHER OUTCOMES:
Blinding effectiveness evaluation | At 2 weeks after the start of the intervention
  The participants, evaluators and those who apply the intervention will be asked if they know the research group to which the study subject belongs through a questionnaire prepared by one of the principal investigators.

CONTACTS AND LOCATIONS:
Overall Officials: Aníbal Báez-Suárez, PhD, Principal Investigator — University of Las Palmas de Gran Canaria
Locations (1):
- Aníbal Báez-Suárez, Las Palmas de Gran Canaria, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wein AJ, Rovner ES. Definition and epidemiology of overactive bladder. Urology. 2002 Nov;60(5 Suppl 1):7-12; discussion 12. doi: 10.1016/s0090-4295(02)01784-3. PMID 12493342
- [Result] Tubaro A. Defining overactive bladder: epidemiology and burden of disease. Urology. 2004 Dec;64(6 Suppl 1):2-6. doi: 10.1016/j.urology.2004.10.047. PMID 15621220
- [Result] Eapen RS, Radomski SB. Review of the epidemiology of overactive bladder. Res Rep Urol. 2016 Jun 6;8:71-6. doi: 10.2147/RRU.S102441. eCollection 2016. PMID 27350947
- [Result] Irwin DE, Milsom I, Hunskaar S, Reilly K, Kopp Z, Herschorn S, Coyne K, Kelleher C, Hampel C, Artibani W, Abrams P. Population-based survey of urinary incontinence, overactive bladder, and other lower urinary tract symptoms in five countries: results of the EPIC study. Eur Urol. 2006 Dec;50(6):1306-14; discussion 1314-5. doi: 10.1016/j.eururo.2006.09.019. Epub 2006 Oct 2. PMID 17049716
- [Result] Ganz ML, Smalarz AM, Krupski TL, Anger JT, Hu JC, Wittrup-Jensen KU, Pashos CL. Economic costs of overactive bladder in the United States. Urology. 2010 Mar;75(3):526-32, 532.e1-18. doi: 10.1016/j.urology.2009.06.096. Epub 2009 Dec 29. PMID 20035977
- [Result] Lightner DJ, Gomelsky A, Souter L, Vasavada SP. Diagnosis and Treatment of Overactive Bladder (Non-Neurogenic) in Adults: AUA/SUFU Guideline Amendment 2019. J Urol. 2019 Sep;202(3):558-563. doi: 10.1097/JU.0000000000000309. Epub 2019 Aug 8. PMID 31039103
- [Result] de Groat WC, Tai C. Impact of Bioelectronic Medicine on the Neural Regulation of Pelvic Visceral Function. Bioelectron Med. 2015 Jan 22;2015:25-36. PMID 26491706
- [Result] Jaqua K, Powell CR. Where Are We Headed with Neuromodulation for Overactive Bladder? Curr Urol Rep. 2017 Aug;18(8):59. doi: 10.1007/s11934-017-0711-x. PMID 28656519
- [Result] Janssen DA, Martens FM, de Wall LL, van Breda HM, Heesakkers JP. Clinical utility of neurostimulation devices in the treatment of overactive bladder: current perspectives. Med Devices (Auckl). 2017 Jun 1;10:109-122. doi: 10.2147/MDER.S115678. eCollection 2017. PMID 28615976
- [Result] Timmermans L, Falez F, Melot C, Wespes E. Validation of use of the International Consultation on Incontinence Questionnaire-Urinary Incontinence-Short Form (ICIQ-UI-SF) for impairment rating: a transversal retrospective study of 120 patients. Neurourol Urodyn. 2013 Sep;32(7):974-9. doi: 10.1002/nau.22363. Epub 2012 Dec 31. PMID 23281067